CLINICAL TRIAL: NCT03883165
Title: How do the Neck Muscles Influence Head Acceleration During Sport-associated Impact Events in High School Athletes?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, James Eckner, Associate Professor of Physical Medicine and Rehabilitation, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HUM00152807; 1R01HD093733-01A1 (NIH)
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Sport-related Concussion; Brain Concussion; Healthy
Keywords: Concussion; Contact sport; Collision sport; Neck strengthening; Soccer; Head Acceleration
MeSH Terms: conditions — Brain Concussion | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither subjects nor the study team members responsible for performing the laboratory- or radiology-based assessment will be informed of group allocation status, although subjects will be aware of whether or not they are performing neck strengthening exercises during their exercise sessions. Subjects will be instructed not to reveal their group status during subsequent assessment sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-intensity neck strengthening group (Experimental)
  Interventions: Other: high-intensity neck strengthening
- Control group (Other)
  Interventions: Other: Control group

INTERVENTIONS:
Other: high-intensity neck strengthening — All subjects will exercise 2 days per week for 12 weeks under the direct supervision of a study-assigned strength coach with a minimum of 1 day of rest between exercise sessions.
  Participants will perform a standardized set of general resistance exercises targeting the chest, shoulders, back, upper and lower extremities, and core. Additionally, they will also perform a higher number of repetitions of manual resistance neck strengthening exercises in sagittal plane flexion and extension, coronal plane lateral flexion in both directions, and axial plane rotation in both directions,as well as dumbbell shoulder shrugs.
  Arms: high-intensity neck strengthening group
Other: Control group — All subjects will exercise 2 days per week for 12 weeks under the direct supervision of a study-assigned strength coach with a minimum of 1 day of rest between exercise sessions.
  Participants will perform a standardized set of general resistance exercises targeting only the chest, shoulders, back, upper and lower extremities, and core, without resistance exercises specifically targeting the neck.
  Arms: Control group

SUMMARY:
Sport-related concussion is a common and serious injury that can affect athletes of all ages in any sport. The purpose of this project is to study the effect of a 12-week manual resistance neck strengthening exercise program on participants' neck size and strength and how their heads and necks move during simulated sport-associated tasks. This study will help determine if greater neck strength may lower an athlete's risk of sport-related concussion. Each healthy male and female soccer athlete between the ages of 13-19 enrolled in the study will participate for approximately four months. Study participation includes routine visits with various assessments (i.e. certain body measurements, magnetic resonance imaging, ultrasound) in addition to the strengthening exercise program.

DETAILED DESCRIPTION:
This study was updated to remove the low-volume group and the amendment was approved 3/29/2023 at the Institutional Review Board. This change to remove the low-volume exercise group was due to reduced enrollment numbers following the Corona Virus Disease (COVID) Pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form, or assent form with parental consent for minors
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Participated in a soccer team, club, or other soccer program/organization within the preceding 2 years
* Be willing to adhere to the assigned exercise regimen

Exclusion Criteria:

* Prior history of trauma-induced neck injury of sufficient severity to require treatment by a medical provider within 30 days of injury or to limit sport participation for > 1 day (note: having received routine chiropractic treatment in the absence of a recent traumatic injury to the neck will not be considered to meet this criterion)
* Any prior history of whiplash injury, stinger/burner, or cervical radiculopathy diagnosed by a medical provider
* Any prior history of bone, disk, neural, or ligamentous abnormality identified on cervical spine medical imaging performed for any reason that is felt by the PI (or designee) to present a risk to study participation
* Any prior history of surgery involving the cervical spine (note: having undergone non-spine surgery to the soft tissue structures in the neck will not necessarily exclude participation, but will be considered on a case-by-case basis by the PI, or his designee, with consultation from the performing surgeon when deemed appropriate)
* Self-report of moderate or severe neck pain (rated as 5 or greater on a 10-point pain scale) lasting > 1 day in the previous 6 months that required any evaluation or treatment by a medical provider or that limited sport participation for > 1 day (note: having received routine chiropractic treatment in the absence of moderate-severe neck pain will not be considered to meet this criterion)
* Self-report of low back pain (any severity) associated with morning stiffness occurring 30 days or more in the previous 3 months.
* Prior episode(s) of unexplained upper extremity numbness, tingling, or weakness suspicious to the PI, or designee, for a stinger/burner or cervical radiculopathy in the last 3 years
* Prior history of concussion in the previous 6 months diagnosed by a medical provider or suspected by the subject, or the parent/guardian of a minor (if no medical evaluation was sought), or any diagnosed/suspected concussion without full recovery and clearance to resume unrestricted sport participation.
* Personal history of migraine headaches within the previous 3 years diagnosed by a medical provider, with one or more headache episodes, or requiring treatment.
* Personal history of anxiety disorder diagnosed by a medical provider that has either been difficult to control, affected daily function, or required treatment with medication or counseling within the previous 3 years.
* Parental/guardian known history of anxiety disorder diagnosed by a medical provider that has either been difficult to control, affected daily function, or required treatment with medication or counseling within the previous 3 years.
* Prior personal of any of the following or known family history of the following medical conditions known to be associated with atlanto-axial instability diagnosed by a medical provider: parental history of Down Syndrome, Ehlers-Danlos Syndrome, or Marfan syndrome; parental, or sibling history of rheumatoid arthritis/other systemic inflammatory disease with joint involvement or mucopolysaccharidosis
* Known exposure to or infection with head lice in the previous 30 days
* Known or suspected pregnancy (for females)
* Serious allergic reaction to nickel/metal jewelry
* Any contraindication to MRI scanning
* Presence of significant abnormality on a standardized screening neurological and musculoskeletal physical examination
* Prior participation in a resistance exercise training program including exercises specifically intended to target the neck muscles within 3 months of enrollment, or intention to begin participating in such an exercise program outside of the study protocol during the upcoming 12-week study period
* Unable to speak and understand English

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2024-06-08 (Actual); Study Completion 2024-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James T Eckner, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eckner JT, Goshtasbi A, Curtis K, Kapshai A, Myyra E, Franco LM, Favre M, Jacobson JA, Ashton-Miller JA. Feasibility and Effect of Cervical Resistance Training on Head Kinematics in Youth Athletes: A Pilot Study. Am J Phys Med Rehabil. 2018 Apr;97(4):292-297. doi: 10.1097/PHM.0000000000000843. PMID 29557889
- [Background] Eckner JT, Oh YK, Joshi MS, Richardson JK, Ashton-Miller JA. Effect of neck muscle strength and anticipatory cervical muscle activation on the kinematic response of the head to impulsive loads. Am J Sports Med. 2014 Mar;42(3):566-76. doi: 10.1177/0363546513517869. Epub 2014 Jan 31. PMID 24488820
- See also: Related Info — https://journals.lww.com/ajpmr/abstract/2018/04000/feasibility_and_effect_of_cervical_resistance.10.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment indicates participants who consented. Prior to randomization 5 participants were lost (2 withdrew, 2 lost to follow-up and 1 no longer eligible).
Period: Overall Study
Arm/Group | Control Group | High-intensity Neck Strengthening Group
Started (Started indicates participants who were randomized after completing their baseline evaluation.) | 24 | 19
Follow-Up Visit 1 | 21 | 19
Follow-Up Visit 2 | 21 | 18
Follow-Up Visit 3 | 20 | 16
Completed | 20 | 16
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-intensity Neck Strengthening Group | Control Group | Total
Number analyzed (Participants) | 19 | 24 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.11 (1.10) | 15.75 (1.54) | 15.47 (1.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 11 | 16 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 16 | 22 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 19 | 34
  More than one race | 3 | 2 | 5
  Other | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 24 | 43

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Net Head Acceleration vs. Time Curve During Direct Loading, With Anticipatory Bracing - Linear Motion.
Description: The linear component of head acceleration was measured with a sensor attached to the head, while a device applied force to the head. The data is reported where higher values represent greater acceleration per amount of force delivered (zero represents no acceleration and greater numbers higher acceleration).
Time Frame: 4 weeks, 8 weeks, 12 weeks
Population: For the high-intensity group 3 subjects withdrew from follow-up visit 1 to Follow-Up Visit 3. For the control group 4 subjects withdrew from the baseline visit to follow-up visit 3.
Measure: Mean (Standard Deviation); unit: meters per second per joule
Arm/Group | High-intensity Neck Strengthening Group | Control Group
Number analyzed (Participants) | 19 | 24
meters per second per joule
  Baseline | .895 (.378) | 1.069 (.501)
  Follow-Up Visit 1 (4 weeks): number analyzed (Participants) | 19 | 21
  Follow-Up Visit 1 (4 weeks) | .873 (.398) | .903 (.491)
  Follow-Up Visit 2 (8 weeks): number analyzed (Participants) | 18 | 21
  Follow-Up Visit 2 (8 weeks) | .893 (.44) | .937 (.404)
  Follow-Up Visit 3 (12 weeks): number analyzed (Participants) | 16 | 20
  Follow-Up Visit 3 (12 weeks) | .839 (.392) | .793 (.386)

2. Primary Outcome: Mean Area Under the Net Head Acceleration vs. Time Curve During Direct Loading, With Anticipatory Bracing - Angular Motion.
Description: The angular component of head acceleration was measured with a sensor attached to the head, while a device applied force to the head. The data is reported where higher values represent greater acceleration per amount of force delivered (zero represents no acceleration and greater numbers higher acceleration).
Time Frame: 4 weeks, 8 weeks, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: radians per second per joule
Arm/Group | High-intensity Neck Strengthening Group | Control Group
Number analyzed (Participants) | 19 | 24
radians per second per joule
  Baseline | .057 (.040) | .069 (.047)
  Follow-Up Visit 1 (4 weeks): number analyzed (Participants) | 19 | 21
  Follow-Up Visit 1 (4 weeks) | .054 (.036) | .058 (.043)
  Follow-Up Visit 2 (8 weeks): number analyzed (Participants) | 18 | 21
  Follow-Up Visit 2 (8 weeks) | .056 (.037) | .063 (.039)
  Follow-Up Visit 3 (12 weeks): number analyzed (Participants) | 16 | 20
  Follow-Up Visit 3 (12 weeks) | .05 (.039) | .049 (.035)

3. Secondary Outcome: Mean Area Under the Net Head Acceleration vs. Time Curve During Indirect Loading, With Anticipatory Bracing - Linear Motion.
Description: The linear component of head acceleration was measured with a sensor attached to the head, while a simulated body check was administered. The data is reported where higher values represent greater acceleration (zero represents no acceleration and greater numbers higher acceleration).
Time Frame: 4 weeks, 8 weeks, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | High-intensity Neck Strengthening Group | Control Group
Number analyzed (Participants) | 19 | 24
meters per second
  Baseline | 1.007 (0.417) | 1.105 (0.432)
  Follow-Up Visit 1 (4 weeks): number analyzed (Participants) | 19 | 21
  Follow-Up Visit 1 (4 weeks) | 1.007 (0.418) | 0.943 (0.403)
  Follow-Up Visit 2 (8 weeks): number analyzed (Participants) | 18 | 21
  Follow-Up Visit 2 (8 weeks) | 0.999 (0.367) | 0.973 (0.323)
  Follow-Up Visit 3 (12 weeks): number analyzed (Participants) | 16 | 20
  Follow-Up Visit 3 (12 weeks) | 0.938 (0.367) | 1.007 (0.397)

4. Secondary Outcome: Mean Area Under the Net Head Acceleration vs. Time Curve During Indirect Loading, With Anticipatory Bracing - Angular Motion.
Description: The angular component of head acceleration was measured with a sensor attached to the head, while a simulated body check was administered. The data is reported where higher values represent greater acceleration (zero represents no acceleration and greater numbers higher acceleration).
Time Frame: 4 weeks, 8 weeks, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: radians per second
Arm/Group | High-intensity Neck Strengthening Group | Control Group
Number analyzed (Participants) | 19 | 24
radians per second
  Baseline | 0.020 (0.010) | 0.020 (0.008)
  Follow-Up Visit 1 (4 weeks): number analyzed (Participants) | 19 | 21
  Follow-Up Visit 1 (4 weeks) | 0.02 (0.011) | 0.018 (0.01)
  Follow-Up Visit 2 (8 weeks): number analyzed (Participants) | 18 | 21
  Follow-Up Visit 2 (8 weeks) | 0.02 (0.008) | 0.019 (0.008)
  Follow-Up Visit 3 (12 weeks): number analyzed (Participants) | 16 | 20
  Follow-Up Visit 3 (12 weeks) | 0.019 (0.009) | 0.019 (0.009)

ADVERSE EVENTS:
Time Frame: Up to four months
Arm/Group | Control Group | High-intensity Neck Strengthening Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/24 | 1/19
Other Adverse Events (participants affected / at risk) | 15/24 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=24) | High-intensity Neck Strengthening Group (N=19)
Nausea (Gastrointestinal disorders) | 0 | 1 — Nausea requiring ER visit, but not hospital admittance.
vomiting (Gastrointestinal disorders) | 0 | 1 — Vomiting requiring ER visit, but not hospital admittance.
Diarrhea (Gastrointestinal disorders) | 0 | 1 — Diarrhea requiring ER visit, but not hospital admittance.
conjunctivitis (Eye disorders) | 1 | 0 — Conjunctivitis requiring ER visit, but not hospital admittance.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=24) | High-intensity Neck Strengthening Group (N=19)
Back pain (General disorders) | 2 | 0
Minor hand injury (Injury, poisoning and procedural complications) | 1 | 0
Headache (General disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Wisdom teeth removal surgery (Surgical and medical procedures) | 2 | 0
Sore throat (General disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Calf cramping (Musculoskeletal and connective tissue disorders) | 1 | 0
Bilateral nerve pain in arms (Nervous system disorders) | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Ankle injury (Injury, poisoning and procedural complications) | 1 | 3
Cold/flu symptoms (Infections and infestations) | 1 | 0
Hip pain (Musculoskeletal and connective tissue disorders) | 1 | 1
COVID (Infections and infestations) | 0 | 1
Knee discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Back spasms (General disorders) | 0 | 1
Fatigue after extensive exertion (General disorders) | 1 | 0
Neck pain (General disorders) | 0 | 1
Knee injury (Injury, poisoning and procedural complications) | 1 | 1
Toe injury (Injury, poisoning and procedural complications) | 1 | 0
Suspected concussion (Injury, poisoning and procedural complications) | 1 | 1
Confirmed concussion (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT03883165/Prot_SAP_001.pdf
  • Informed Consent Form (2023-12-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT03883165/ICF_000.pdf